CLINICAL TRIAL: NCT01363739
Title: Prospective Evaluation of -1498 c/t VEGF Polymorphism in the Prediction of Benefit From First-line Folfiri Plus Bevacizumab in Metastatic Colorectal Cancer Patients
Brief Title: Evaluation of VEGF Polymorphism as Predictive Factor in Metastatic Colorectal Cancer Treated With Folfiri Plus Bevacizumab
Acronym: PROVETTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Alfredo Falcone, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: 3108
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: VEGF polymorphism Bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
-1498C/T VEGF polymorphism, as suggested by a recent retrospective analysis, seems to have a role in predicting the efficacy of Bevacizumab plus FOLFIRI in first-line treatment of metastatic colorectal cancer patients. The present study aims to prospectively evaluate the predictive role of this polymorphism in metastatic colorectal patients receiving the same treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal adenocarcinoma;
* Measurable metastatic disease according to RECIST criteria;
* Patients receiving BV plus FOLFIRI as first-line treatment;
* Written informed consent;
* Availability of blood samples for genetic analysis.-

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Metastatic colorectal cancer patients receiving FOLFIRI plu Bevacizumab as first-line treatment
Sampling Method: Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2009-04

PRIMARY OUTCOMES:
Progression-Free Survival
  Progression free survival (PFS) is defined as time from study entry until progression of disease (according to RECIST 1.1) or death from any cause. Patients who are alive without having progressed at the end of the study will be censored at their last radiological assessment

SECONDARY OUTCOMES:
Response Rate
  Response Rate (RR) is defined as the fraction of treated patients who achieve a response as defined according to Response Evaluation Criteria in Solid Tumors (RECIST)
Overal survival
  Overall survival (OS) is defined as the time from study entry until death from any cause. Patients who are alive at the end of the study will be censored at that point

CONTACTS AND LOCATIONS:
Locations (1):
- Polo Oncologico Azienda Ospedaliero, Universitaria Pisana, Pisa, Pisa, Italy